CLINICAL TRIAL: NCT03553771
Title: A French, Multicenter, Prospective, Observational, "Real Life" Assessment of the Safety and Efficacy of the Low Profile Visualized Intraluminal Support (LVIS and LVIS JR) Devices in the Treatment of Intracranial Aneurysms
Brief Title: Safety and Efficacy of the LVIS and LVIS JR Devices in the Endovascular Treatment of Intracranial Aneurysms
Status: Completed | Type: Observational
Sponsor: Microvention-Terumo, Inc. (Industry)
Collaborators: Clinact (Other)
Responsible Party: Sponsor
Other Study IDs: LEPI
Record Dates: First submitted 2018-05-16; First posted 2018-06-12 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Intracranial Aneurysm
Keywords: aneurysm; endovascular
MeSH Terms: conditions — Intracranial Aneurysm; Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: LVIS and LVIS JR — Braided coil assist stents used for aneurysm embolization
  Other Names: Low Profile Visualized Intraluminal Support

SUMMARY:
A French, multicenter, prospective, observational, "real life" assessment of the safety and efficacy of LVIS and LVIS JR devices in the treatment of intracranial aneurysms

DETAILED DESCRIPTION:
This is a multicenter observational study. Treatment and follow-up visits will be done as per standard of care.

The purpose of this study is to collect data on safety of the devices used since the French reimbursement.

130 patients will be enrolled over an 18-month recruitment period. All patients will be followed for at least 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient with an intracranial aneurysm for which an endovascular treatment is indicated with the device LVIS or LVIS JR, either scheduled or emergency (" Bail-out stenting ")
* Patient or patient's legally authorized representative has been informed about the study and does not oppose the collection of his/her personal data

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with ruptured or not ruptured intracranial aneurysms treated with LVIS or LVIS Jr stent
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2018-02-07 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Mortality Rate | 1 year
Morbidity Rate | 1 year
  Number of adverse events with clinical impact related to the procedure and/or the device

SECONDARY OUTCOMES:
Clinical effectiveness | 1 year
  Number of patients with mRS>2
Anatomical effectiveness | 1 year
  Number of patients with complete occlusion of the treated aneurysm
Retreatment rate | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Michel Piotin, MD, Principal Investigator — Fondation Rothschild, Paris, France; Charbel Mounayer, Prof., Principal Investigator — CHU de Limoges, France
Locations (20):
- France (20):
  - CHU Pellgrin, Bordeaux
  - CHU Caen, Caen
  - CHU Gabriel Montpied, Clermont-Ferrand
  - CHU Michallon, Grenoble
  - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - CHU Limoges, Limoges
  - Hôpital Clairval, Marseille
  - Hôpital de la Timone, Marseille
  - Hôpital Gui de Chauliac, Montpellier
  - Hôpital Central de Nancy, Nancy
  - Hôpital Pasteur 2, Nice
  - Hôpital Lariboisière, Paris
  - Hôpital Pitié-Salpêtrière, Paris
  - La Fondation Rothschild, Paris
  - Hôpital Maison Blanche, Reims
  - Hôpital Nord, Saint-Etienne
  - Hôpital Foch, Suresnes
  - Hôpital d'instruction des Armées Saint-Anne, Toulon
  - Hôpital Purpan, Toulouse
  - Hôpital Bretonneau, Tours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Forestier G, Piotin M, Chau Y, Derelle AL, Brunel H, Aggour M, Saleme S, Levrier O, Pierot L, Barreau X, Boubagra K, Janot K, Barbier C, Clarencon F, Chabert E, Spelle L, Arteaga C, Consoli A, Machi P, Blanc R, Rodesch G, Cortese J, Sourour N, Herbreteau D, Heck O, Soize S, Marnat G, Rouchaud A, Anxionnat R, Sedat J, Mounayer C; LEPI investigators. Safety and effectiveness of the LVIS and LVIS Jr devices for the treatment of intracranial aneurysms: Final results of the LEPI multicenter cohort study. J Neuroradiol. 2024 May;51(3):242-248. doi: 10.1016/j.neurad.2023.10.007. Epub 2023 Oct 17. PMID 37858720
- See also: Safety and effectiveness of the LVIS and LVIS Jr devices for the treatment of intracranial aneurysms: Final results of the LEPI multicenter cohort study — https://pubmed.ncbi.nlm.nih.gov/37858720/